CLINICAL TRIAL: NCT02690337
Title: Phase 1, Open-label Study to Assess the Safety, Tolerability, and Pharmacokinetics of DS-1123a in Subjects With Advanced Solid Tumors
Brief Title: Study of DS-1123a in Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS1123-A-J101
Record Dates: First submitted 2016-02-04; First posted 2016-02-24 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-01

CONDITIONS: Advanced Solid Malignant Tumors
Keywords: Advanced solid malignant tumors; phase 1; oncology; refractory; no standard treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DS-1123 (Experimental): This study will follow a modified Continual Reassessment Method (mCRM) + Escalation with Overdose Control (EWOC),design with a starting intravenous (IV) dose of 0.1 mg/kg.
  Interventions: Drug: DS-1123

INTERVENTIONS:
Drug: DS-1123 — starting intravenous (IV) dose of 0.1 mg/kg.

SUMMARY:
This is an open-label study to evaluate the safety, tolerability, and pharmacokinetics of DS-1123a in Japanese subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor that is refractory to standard treatment, or for which no standard treatment is available.
* Eastern Cooperative Oncology Group performance status (PS) of 0 or 1.

Exclusion Criteria:

* Have any of the following concomitant disease or had the history of having following disease within 6 months before enrollment:

  • Cardiac failure (NYHA ≥ ClassIII), myocardial infarction, cerebral infarction, unstable angina, arrhythmia requiring treatment, coronary-artery/peripheral artery bypass surgery, cerebrovascular disease, pulmonary thromboembolism, deep-vein thrombosis or clinically severe thromboembolic event, or clinically severe pulmonary disease (eg, interstitial pneumonia, pulmonary fibrosis, radiation pneumonia, drug induced pneumonia),
* Severe or uncontrolled concomitant disease.
* Clinically active brain metastases defined as symptomatic or requiring treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | Cycles 1, 2 : Days 1,2, 4, 8, 15
Number and severity of treatment emergent adverse events (TEAEs) | Day 1 to Day 31
Time of maximum concentration (Tmax) | Cycles 1, 2: Days 1,2, 4, 8, 15
Elimination rate constant (Kel) | Cycles 1, 2: Days 1,2, 4, 8, 15
area under the curve AUClast | Cycles 1, 2: Days 1,2, 4, 8, 15
  pharmacokinetics profile
Area under the curve (AUCtau) | Cycles 1, 2: Days 1,2, 4, 8, 15
Area under the curve (AUCinf) | Cycles 1, 2: Days 1,2, 4, 8, 15
Half-life (T1/2) | Cycles 1, 2: Days 1,2, 4, 8, 15
Drug clearance (CL) | Cycles 1, 2: Days 1,2, 4, 8, 15
Volume of distribution (Vz) | Cycles 1, 2: Days 1,2, 4, 8, 15
Mean residence time (MRTinf) | Cycles 1, 2: Days 1,2, 4, 8, 15

SECONDARY OUTCOMES:
DS-1123a antibody | Cycle 1: Days 1,15; Cycles 2: Day 1; Stop date, final follow-up date
  DS-1123a antibody on Cycle 1: Days 1,15; Cycles 2 and on: Day 1, Stop date, final follow-up date
Change in Cytokines expression | Cycle 1: Days 1, 2, 15, 16; Cycle 2: Days 1, 2
  Change in DS-1123a biomarkers Cytokines expression on Cycle 1: Days 1, 2, 15, 16; Cycle 2: Days 1, 2

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/